CLINICAL TRIAL: NCT03245697
Title: Breast Milk Composition: Interindividual Variations and Dietary Factors in Galicia
Status: Completed | Type: Observational
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, PATRICIA REGAL, Professor and PhD researcher, University of Santiago de Compostela
Other Study IDs: 2016-CL045
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Milk, Human
Keywords: breast milk; composition; Galicia; diet; lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lactating mothers: Lactating mothers recruited in Galicia (NW Spain)

SUMMARY:
Human milk is not a uniform body fluid, but quite the opposite, its composition changes continuously adapting to the requirements of the newborn. It can be considered as the gold standard for infants' nutrition and exclusive breastfeeding is recommended by the WHO during the first months of life. Additionally, its composition should be used as reference or guidance for defining optimal nutrient intakes for infants that cannot be fully breastfed. In that connection, the nutritional status and dietary habits/patterns of the mother, along with certain genetic traits, exert also influence over breast milk. Considering all these facts, and their great impact on (present and future) infant health, detailed information of breast milk composition is required for specific populations, covering as many factors, elements and nutrients as possible.

In the present observational study, research is focused on breast milk in northwestern Spain, more precisely Galicia. In this context, the obtained data will serve to define the nutritional characteristics of breast milk from Galician women (interindividual variation), while at the same time evaluating the existence of specific features related to their particular diet (dietary factors), the Southern European Atlantic Diet (SEAD). All the variables measured in this research project will be related with breast milk composition. Expected primary outcomes can be divided as follows: fatty acid profiles, mineral composition, essential amino acid profiles, microbiota and steroid hormones. The key influencing factors taken into account are: lactation characteristics and maternal diet.

Recruitment of participants is based on all the following criteria, with no exceptions: female, living in Galicia, lactating, > 18 years old, volunteer participation, written informed consent and agreement to complete questionnaires about lactation, diet and other socio-demographic factors. Samples are collected by participants, and stored at the University of Santiago de Compostela under a coded system so that it is impossible to identify the donor from whom the sample comes, with the exception of the investigators. The project is adhered to the principles of the Helsinki Declaration. Participants are allowed to withdraw their consent at any moment of the study.

ELIGIBILITY:
Inclusion Criteria:

* female
* lactating
* living in Galicia
* voluntary participation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Lactating mothers
Study Population: Lactating/nursing women living in northwestern Spain (Galicia)
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Fatty acid profile of breast milk in Galicia | 2016
  Fatty acid profile of breast milk collected from lactating women in Galicia, at different points postpartum; discussion on diet influence.

CONTACTS AND LOCATIONS:
Overall Officials: PATRICIA REGAL, PhD, Principal Investigator — University of Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Undecided